CLINICAL TRIAL: NCT01340469
Title: Nosocomial Infections and Necrotizing Enterocolitis in Preterm Neonates Treated With Lactobacillus Acidophilus and Bifidobacterium Infantis in An Intensive Care Unit : A Randomized Controlled Study
Brief Title: Effect of Oral Probiotic Supplementation on The Rate of Hospital Acquired Infection and Necrotizing Enterocolitis in Preterm Very Low Birth Weight Infants
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: King Chulalongkorn Memorial Hospital (Other)
Responsible Party: Santi Punnahitananda, Faculty of Medicine Chulalongkorn University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 076/2003
Record Dates: First submitted 2011-04-19; First posted 2011-04-22 (Estimated); Last update posted 2011-04-22 (Estimated); Status verified 2011-03

CONDITIONS: Nosocomial Infection; Necrotizing Enterocolitis
Keywords: nosocomial infections; necrotizing enterocolitis; preterm infants; ver low birth weight; probiotics
MeSH Terms: conditions — Cross Infection; Enterocolitis, Necrotizing | interventions — Probiotics

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- study (Active Comparator): Probiotics supplementation .
  Interventions: Biological: probiotics
- control (Placebo Comparator): The control group received daily placebo liquid .
  Interventions: Biological: probiotics

INTERVENTIONS:
Biological: probiotics — Daily enteral probiotic supplementation (live Lactobacillus acidophilus and Bifidobacterium infantis) at a dose of 2.5 x 108 CFU of each strain once a day.The supplementation was started on the first day of enteral feeding and continued for at least 28 days or until discharge. The study drug was in liquid form and mixed with breast milk or formula before given to the infants. The preparation was made on a daily basis by one person who was not involved in the care of the infants.
  Other Names: Infloran (Swiss Berna)

SUMMARY:
The purpose of this study is to determine whether oral probiotic supplementation could reduce the incidence of nosocomial infections in preterm infants.

DETAILED DESCRIPTION:
There are growing numbers of evidence indicating the beneficial effects of normal enteric flora (probiotics) with regard to the host defense against infection. In vitro and in vivo studies have shown that probiotics such as lactobacilli and bifidobacteria have inhibitory effects on other pathogenic bacteria.This evidence, along with the results of recent clinical studies, has demonstrated the beneficial effects of probiotics in the prevention of NEC in VLBW infants.However, most of the studies reported nosocomial infection as a secondary outcome and the findings were controversial regarding probiotics efficacy in preventing nosocomial infections. There is only one study that was aimed to investigate effects of probiotic on the incidence of nosocomial infection.

Given the potential benefit of probiotics against infection and the lack of clinical studies in this regard, we conducted a randomized clinical trial to determine whether probiotic supplementation (in the form of Lactobacillus acidophilus and Bifidobacterium infantis) could reduce nosocomial infection rate among preterm VLBW infants in a intensive care nursery setting.

ELIGIBILITY:
Inclusion Criteria:

* Very Low Birth Weight (VLBW) preterm infants (Gestational age < 35 weeks , BW < 1500 g ) admitted to the NICU who survived the first 3 days of life

Exclusion Criteria:

* Infants with chromosome abnormality or severe congenital defects, especially gastrointestinal anomalies (e.g. omphalocele, gastroschisis, intestinal obstruction) and infants with unstable hemodynamic status

Ages: 3 Days to 28 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 160 (Estimated)
Dates: Start 2005-01; Primary Completion 2008-03 (Actual); Study Completion 2008-06 (Actual)

PRIMARY OUTCOMES:
incidence of nosocomial infections | 28 days or until discharge
  Nosocomial infections , defined as any major infection occurring during the hospitalization, not earlier than 5 days of life.(sepsis, pneumonia, NEC, meningitis, omphalitis, osteomyelitis, soft tissue infection etc.). Sepsis was defined as a clinical syndrome of systemic illness accompanied by positive blood culture.

SECONDARY OUTCOMES:
incidence of necrotizing enterocolitis (NEC) | 28 days or until discharge
  necrotizing enterocolitis (NEC), which was identified and categorized by modified Bell's classification
feeding tolerance | 28 days
  the volume of feeding on day 7,14,21, and 28 of study
time to full enteral feeding | 28 days
  time required to reach full feeding at 150 ml/kg/day

CONTACTS AND LOCATIONS:
Overall Officials: Santi Punnahitananda, M.D., Principal Investigator — Chulalongkorn University
Locations (1):
- Faculty of Medicine Chilalongkorn University, Bangkok, Bangkok, Thailand